CLINICAL TRIAL: NCT04906759
Title: A Meal Delivery and Exercise Intervention to Increase Resilience in Homebound Older Adults
Brief Title: Meal Delivery and Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jessica Lee, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSC-MS-21-0125; 1K23AG072042-01 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Frailty
Keywords: homebound patients; exercise; nutrition
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Meals; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meals plus exercise (Experimental)
  Interventions: Behavioral: Meals plus exercise
- Meals only (Experimental)
  Interventions: Behavioral: Meals only

INTERVENTIONS:
Behavioral: Meals plus exercise — Participants will receive 12 weeks of a MOW delivery service that will include 2 meals per day during the weekdays with 4 shelf-stable meals at the end of the week. The MOW driver will visit the participants in-person to ask a series of 5 questions about change in health status, joint/muscle injuries, new pain, falls, and poor appetite twice a week. Participants will also will receive an exercise kit from the MOW driver with their first meal delivery which will contain 2 tennis balls, 2 1-pound hand weights, and one towel. Every week, the driver will give the participants a handout containing 3 exercises from the NIA Go4Life Workout-to-Go book that are designed to help with strength/endurance, balance, and flexibility20. The participants will be asked to do the 3 exercises every day, if possible, on their own. Every 4 weeks during the 12-week study period and at 6 months follow up patients will have blood drawn for frailty and inflammatory biomarkers.
  Arms: Meals plus exercise
Behavioral: Meals only — Participants will receive 12 weeks of a MOW delivery service that will include 2 meals per day during the weekdays with 4 shelf-stable meals at the end of the week. The MOW driver will visit the participants in-person to ask a series of 5 questions about change in health status, joint/muscle injuries, new pain, falls, and poor appetite twice a week. they will be asked to continue their usual level of activity.Every 4 weeks during the 12-week study period and at 6 months follow up patients will have blood drawn for frailty and inflammatory biomarkers.
  Arms: Meals only

SUMMARY:
The purpose of this study is to evaluate the effects of a home-based exercise program administered through Meals on wheels (MOW) on gait speed and frailty status and to assess the association between novel serum biomarkers (70 kilodalton heat shock proteins (HSP70),Macrophage Inflammatory Proteins(MIP1b), soluble IL-6 receptor alpha-chain (sIL-6R)) and established but non-specific frailty biomarkers (Interleukin 6 (IL-6), C-reactive protein (CRP), Tumor necrosis factor (TNF-α)) in frail and prefrail homebound older adults before and after the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* homebound (normally unable to leave the home unassisted)
* frail or prefrail by The Fried Frailty Phenotype (FFP)
* medically stable

Exclusion Criteria:

* robust by FFP
* have Mini-Cog score <3 and/or are unable to follow instructions
* have a pre-diagnosed terminal illness
* unable to ambulate
* unable to use their upper extremities, and/or are already participating in physician-prescribed physical therapy or occupational therapy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in gait speed | 4 weeks,8 weeks,12 weeks from baseline
  this is the time one takes to walk a specified distance on level surfaces over a short distance and is measured in meters/second
Change in total FFP score as assessed by the Fried Frailty Phenotype (FFP) screening test | 4 weeks,8 weeks,12 weeks from baseline
  Score from 0(not frail),1-2(pre frail) and 3-5(frail)
Change in measure of HSP70 (ng/mL) expression | 4 weeks,8 weeks,12 weeks from baseline
Change in Measure of MIP-1β (pg/mL) expression | 4 weeks,8 weeks,12 weeks from baseline
Change in Measure of sIL-6R (pg/mL) expression | 4 weeks,8 weeks,12 weeks from baseline

SECONDARY OUTCOMES:
Change in overall frailty status as assessed by the Fried Frailty Phenotype (FFP) screening test | 4 weeks,8 weeks,12 weeks from baseline
  The FFP defines frailty as having 3 or more characteristics of unintentional weight loss, fatigue, decreased physical activity, weakness, and slowness.Those who have 1 or 2 characteristics are considered pre frail, while those who have no characteristics are robust.
Change in grip strength | 4 weeks,8 weeks,12 weeks from baseline
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles .This is measured by using a dynamometer which will be squeezed by the participant 3 times in each hand.The force is measured in kilograms.
Change in daily average steps from the activity tracker | 4 weeks,8 weeks,12 weeks from baseline
Number of patients that required emergency room visits | 6 months post baseline visit
Number of patients that required hospitalization | 6 months post baseline visit
Change in activities of daily living as measured by the Katz Index of Independence in Activities of Daily Living | 4 weeks,8 weeks,12 weeks from baseline
  This consists of 6 questions and each is scored form 0(patient is very dependent)-6(patient is independent)
Change in instrumental activities of daily living as measured by the LAWTON - BRODY INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE (I.A.D.L.) | 4 weeks,8 weeks,12 weeks from baseline
  This consists of 8 questions and each has a summary score range from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Change in loneliness as assessed by the UCLA Loneliness Scale (ULS) | 4 weeks,8 weeks,12 weeks from baseline
  This questionnaire consists of 20 questions and each is answered from 1(never)-4(always) for a total score ranging form 20-80
Social network as assessed by the LUBBEN SOCIAL NETWORK SCALE - 18 (LSNS-18) | 4 weeks,8 weeks,12 weeks from baseline
  LSNS-R total score is an equally weighted sum of twelve items. Scores range from 0 to 90, a higher number indicating a better outcome
change in measure of IL-6 (pg/mL) expression | 4 weeks,8 weeks,12 weeks from baseline
Change in measures of CRP (ng/mL) expression | 4 weeks,8 weeks,12 weeks from baseline
Change in measures of TNF-α (pg/mL) expression | 4 weeks,8 weeks,12 weeks from baseline
Change in measures of microbiome (fecal sample) expression | 4 weeks,8 weeks,12 weeks from baseline
change in IL-6 (pg/mL) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline
change in CRP (ng/mL) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline
change in TNF-α (pg/mL) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline
change in HSP70 (ng/mL) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline
change in MIP-1β (pg/mL) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline
change in sIL-6R (pg/mL) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline
change in microbiome (fecal sample) as measured by the frailty status | 4 weeks,8 weeks,12 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lee, MD,MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No